CLINICAL TRIAL: NCT06816537
Title: The Effect of Low-level Laser Therapy to Reduce Pain Caused by Orthodontic Separators: A Randomized, Double-blind Place-bo-controlled, Split-mouth Study
Acronym: SZTEDENT-laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Melinda Madléna, Full professor, Szeged University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: SZTE-DENT-2020-38078-6
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Orthodontic Pain
Keywords: orthodontics; orthodontic pain; low-level laser therapy; LLLT; laser; oral health; mandible
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: randomized, double-blind placebo-controlled (RDBPC) split-mouth study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low level laser therapy (Experimental): A low-level medical gallium-aluminum-arsenide (GaAlAs) diode laser device will used on the 1st permanent molars in the test quadrants, to decrease pain associated with the placement of orthodontic separators
  Interventions: Radiation: Low Level Laser Therapy
- No intervention (Placebo Comparator): The handpiece was also held on the placebo treatment side without laser irradiation (fake irradiation) following the same application protocol as the LLLT treatment side.
  Interventions: Other: No Interventions

INTERVENTIONS:
Radiation: Low Level Laser Therapy — A low-level medical gallium-aluminum-arsenide (GaAlAs) diode laser device will be used on the 1st permanent molars in the test quadrants
  Arms: Low level laser therapy
Other: No Interventions — The handpiece was also held on the placebo treatment side without laser irradiation (fake irradiation) following the same application protocol as the LLLT treatment side.
  Arms: No intervention

SUMMARY:
Thirty-three (n=33) participants from the Department of Orthodontics and Pediatric Dentistry, University of Szeged will be randomly assigned into two groups.

A randomly assigned, split-mouth design will be used to avoid inter-individual biologic variation between patients. First, it will be randomly determined whether the upper or lower jaw would be involved in the study; after choosing the jaw blindly, the actual dental arch in the mouth will further be divided vertically, into right and left halves (quadrants) in each patient. One half will be the experimental side (i.e. the test quadrant) and will receive laser therapy, while the other half will be the placebo side (i.e. placebo quadrant) which will receive no laser, only placebo therapy.

In the experimental group, a low-level medical gallium-aluminum-arsenide (GaAlAs) diode laser device (wavelength 980 nm, power: 100mW, producing 6 J energy), with continuous wave will used on the 1st permanent molars in the test quadrants. Using the split mouth design, patients will receive only a single dose immediately after the placement of orthodontic separators. Specified points in each quadrant will be treated from mesial, central and distal directions on the mucosa both buccally and lingually/palatinally with 10-10 sec for each, altogether for 60 sec, producing 36 J energy per molar. During the placebo treatment session, a similar procedure to that of the laser treatment session will be carried out, but with no laser irradiation. Therefore, to control the patient's pain-related behavior, and to maintain the blinded protocol, the handpiece will also be held on the placebo treatment side without laser irradiation following a similar application protocol.

Patients will be instructed to denote their pain sensation levels (which is expected to be the primary come measure of the study), according to the localization (upper/lower jaw; right/left side) and the given appointments following the treatments: at 0 hours (i.e. within 5 minutes of placing the elastic separators), at 6 hours , at 12 hrs , at 24 hrs , at 48 hrs and at 72 hrs ,after treatment (laser/placebo) in resting position of the mandible (spontaneous pain) and during mastication, on a Visual Analog Scale (VAS), ranging from 0 (no pain) to 100 (severe pain).

DETAILED DESCRIPTION:
After finishing the development of the jaws, effective treatment of orthodontic anomalies needs fixed appliances. During initiation of routine orthodontic treatment with fixed appliances, placing elastic separators is a part of the process to achieve adequate space for orthodontic bands, which may lead to a considerable pain experience. This pain experience is a key barrier to the completion of orthodontic treatment processes, therefore, different approaches have been considered to reduce pain due to orthodontic treatment. Earlier studies have evaluated the effects of low level laser therapy (LLLT) on reducing pain caused by orthodontic elastic separators, however, the reported results are still contradictory: while some investigations supported the notion of analgetic effects, while other studies could not verify it. Therefore, due to the controversial position of LLLT as a treatment modality in orthodontic pain, recent reviews on this topic indicated that further, well-designed randomized controlled trials are needed to clarify the role and usefulness of LLLT in reduction of orthodontic pain.

Therefore, the aim of the present study will be to assess the effect of LLLT in reducing pain following orthodontic elastic separator placement in individuals treated with fixed orthodontic appliances, using a randomized, double-blind placebo-controlled split-mouth study design.

Thirty-three (n=33) participants from the Department of Orthodontics and Pediatric Dentistry, University of Szeged will be randomly assigned into two groups. A randomly assigned, split-mouth design will be used to avoid inter-individual biologic variation between patients. First, it will be randomly determined whether the upper or lower jaw would be involved in the study; after choosing the jaw blindly, the actual dental arch in the mouth will further be divided vertically, into right and left halves (quadrants) in each patient. One half will be the experimental side (i.e. the test quadrant) and will receive laser therapy, while the other half will be the placebo side (i.e. placebo quadrant) which will receive no laser, only placebo therapy.

In the experimental group, a low-level medical gallium-aluminum-arsenide (GaAlAs) diode laser device (wavelength 980 nm, power: 100mW, producing 6 J energy), with continuous wave will used on the 1st permanent molars in the test quadrants. Using the split mouth design, patients will receive only a single dose immediately after the placement of orthodontic separators. Specified points in each quadrant will be treated from mesial, central and distal directions on the mucosa both buccally and lingually/palatinally with 10-10 sec for each, altogether for 60 sec, producing 36 J energy per molar. During the placebo treatment session, a similar procedure to that of the laser treatment session will be carried out, but with no laser irradiation. Therefore, to control the patient's pain-related behavior, and to maintain the blinded protocol, the handpiece will also be held on the placebo treatment side without laser irradiation following a similar application protocol.

Patients will be instructed to denote their pain sensation levels (which is expected to be the primary come measure of the study), according to the localization (upper/lower jaw; right/left side) and the given appointments following the treatments: at 0 hours (i.e. within 5 minutes of placing the elastic separators), at 6 hours , at 12 hrs , at 24 hrs , at 48 hrs and at 72 hrs ,after treatment (laser/placebo) in resting position of the mandible (spontaneous pain) and during mastication, on a Visual Analog Scale (VAS), ranging from 0 (no pain) to 100 (severe pain).

ELIGIBILITY:
Eligible participants of the study are going to be included from the pool of patients at the Department of Orthodontics and Pediatric Dentistry (Faculty of Dentistry, University of Szeged) requiring orthodontic treatment.

Inclusion Criteria:

* individuals aged between 18 and 50 years
* completely erupted second molars without open interproximal contacts of the first molars
* good general health, without the existence of systemic diseases
* adequate oral hygiene and healthy periodontium
* no previous orthodontic treatment

Exclusion Criteria:

* those who did not fulfill the general inclusion criteria
* patients who had undergone prior oral LLLT
* who were using painkillers or other NSAIDs
* those who were consumed tobacco products
* pregnant or lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in the level of pain | At 0 hours (h) (i.e. within 5 minutes of placing the elastic separators), at 6 hours (h) (±30 minutes), at 12 hours (±30 minutes), at 24 hours (±30 minutes), at 48 hours (±30 minutes) and at 72 hours (±30 minutes) after treatment (laser/placebo)
  Patients were instructed to denote their pain sensation levels according to the localization (upper/lower jaw; right/left side) after treatment (laser/placebo) in resting position of the mandible (spontaneous pain) and during mastication, on a Visual Analog Scale (VAS), from 0 (no pain) to 100 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Madléna, Prof. Dr., Principal Investigator — Department of Orthodontics and Pediatric Dentistry, Faculty of Dentistry, University of Szeged
Locations (1):
- Department of Orthodontics and Pediatric Dentistry, Faculty of Dentistry, University of Szeged, Szeged, Csongrád-Csanád, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh LJ. The current status of low level laser therapy in dentistry. Part 1. Soft tissue applications. Aust Dent J. 1997 Aug;42(4):247-54. doi: 10.1111/j.1834-7819.1997.tb00129.x. PMID 9316312
- [Background] Ren C, McGrath C, Yang Y. The effectiveness of low-level diode laser therapy on orthodontic pain management: a systematic review and meta-analysis. Lasers Med Sci. 2015 Sep;30(7):1881-93. doi: 10.1007/s10103-015-1743-4. Epub 2015 Mar 24. PMID 25800534
- [Background] Farzan A, Khaleghi K. The Effectiveness of Low-Level Laser Therapy in Pain Induced by Orthodontic Separator Placement: A Systematic Review. J Lasers Med Sci. 2021 Jun 24;12:e29. doi: 10.34172/jlms.2021.29. eCollection 2021. PMID 34733752
- [Background] Qamruddin I, Alam MK, Fida M, Khan AG. Effect of a single dose of low-level laser therapy on spontaneous and chewing pain caused by elastomeric separators. Am J Orthod Dentofacial Orthop. 2016 Jan;149(1):62-6. doi: 10.1016/j.ajodo.2015.06.024. PMID 26718379
- [Background] Farias RD, Closs LQ, Miguens SA Jr. Evaluation of the use of low-level laser therapy in pain control in orthodontic patients: A randomized split-mouth clinical trial. Angle Orthod. 2016 Mar;86(2):193-8. doi: 10.2319/122214-933.1. Epub 2015 Jul 1. PMID 26132512
- [Background] Eslamian L, Borzabadi-Farahani A, Hassanzadeh-Azhiri A, Badiee MR, Fekrazad R. The effect of 810-nm low-level laser therapy on pain caused by orthodontic elastomeric separators. Lasers Med Sci. 2014 Mar;29(2):559-64. doi: 10.1007/s10103-012-1258-1. Epub 2013 Jan 20. PMID 23334785
- [Background] Nobrega C, da Silva EM, de Macedo CR. Low-level laser therapy for treatment of pain associated with orthodontic elastomeric separator placement: a placebo-controlled randomized double-blind clinical trial. Photomed Laser Surg. 2013 Jan;31(1):10-6. doi: 10.1089/pho.2012.3338. Epub 2012 Nov 15. PMID 23153291
- [Background] Artes-Ribas M, Arnabat-Dominguez J, Puigdollers A. Analgesic effect of a low-level laser therapy (830 nm) in early orthodontic treatment. Lasers Med Sci. 2013 Jan;28(1):335-41. doi: 10.1007/s10103-012-1135-y. Epub 2012 Jul 21. PMID 22814893
- [Background] Xiaoting L, Yin T, Yangxi C. Interventions for pain during fixed orthodontic appliance therapy. A systematic review. Angle Orthod. 2010 Sep;80(5):925-32. doi: 10.2319/010410-10.1. PMID 20578865
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Tortamano A, Lenzi DC, Haddad AC, Bottino MC, Dominguez GC, Vigorito JW. Low-level laser therapy for pain caused by placement of the first orthodontic archwire: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2009 Nov;136(5):662-7. doi: 10.1016/j.ajodo.2008.06.028. PMID 19892282
- [Background] Turhani D, Scheriau M, Kapral D, Benesch T, Jonke E, Bantleon HP. Pain relief by single low-level laser irradiation in orthodontic patients undergoing fixed appliance therapy. Am J Orthod Dentofacial Orthop. 2006 Sep;130(3):371-7. doi: 10.1016/j.ajodo.2005.04.036. PMID 16979496
- [Background] Lim HM, Lew KK, Tay DK. A clinical investigation of the efficacy of low level laser therapy in reducing orthodontic postadjustment pain. Am J Orthod Dentofacial Orthop. 1995 Dec;108(6):614-22. doi: 10.1016/s0889-5406(95)70007-2. PMID 7503039
- [Background] Harazaki M, Isshiki Y. Soft laser irradiation effects on pain reduction in orthodontic treatment. Bull Tokyo Dent Coll. 1997 Nov;38(4):291-5. PMID 9566142
- [Derived] Dezfully AK, Gajdacs M, Pato AE, Karpati K, Madlena M. The Effect of Low-Level Laser Therapy to Reduce Pain Caused by Orthodontic Separators: A Randomized, Double-Blind Placebo-Controlled, Split-Mouth Study. Dent J (Basel). 2025 Apr 22;13(5):181. doi: 10.3390/dj13050181. PMID 40422601